CLINICAL TRIAL: NCT03633357
Title: Translational Validation of 5HT7 Antagonists as a Treatment for Cognitive Impairment in Bipolar Disorder: a Proof of Principle Neuroimaging Study
Brief Title: Imaging 5HT7 Antagonist Effects in Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 240244
Record Dates: First submitted 2018-08-08; First posted 2018-08-16 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Cognitive Impairment
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction | interventions — 3-(4-chlorophenyl)-1,4,5,6,7,8-hexahydro-1-(phenylmethyl)pyrazolo(3,4-d)azepine 2-hydroxy-1,2,3-propanetricarboxylate

STUDY DESIGN:
Intervention Model Description: Crossover, Mechanistic Pharmacological Neuroimaging Study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JNJ-18038683 first (Experimental): One week of JNJ-18038683, followed by one week of Placebo after a two week-washout period,
  Interventions: Drug: JNJ-18038683; Drug: Placebo
- Placebo first (Placebo Comparator): One week of Placebo followed by one week of JNJ-18038683 after a two week-washout period,
  Interventions: Drug: JNJ-18038683; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-18038683 — JNJ-18038683 has been developed by Janssen Pharmaceuticals (Johnson and Johnson), and is a relatively selective high affinity functional 5-HT7 receptor antagonist.
  Participants will take two 10-mg tablets daily, for seven days.
Drug: Placebo — Participants will take two placebo tablets daily, for seven days.

SUMMARY:
The main aim of this research is to examine the potential of 5HT7 antagonists for the treatment of cognitive impairment in bipolar disorder by determining the effect of the 5HT7 antagonist JNJ-18038683 on cognitive and emotional processing related brain activity in cognitively impaired people with bipolar disorder and healthy participants using functional MRI (fMRI). This study is designed to contribute to the rational validation of 5HT7 antagonists as a treatment for cognitive impairment in bipolar disorder and to support the development of clinical trials and further drug development in this area. The study will also examine the effect of 5HT7 antagonism on brain function in healthy participants as this has never been investigated before, and to use as a comparator to determine whether 5HT7 antagonism effects disease specific impairments in task related brain activity and cerebral blood flow.

DETAILED DESCRIPTION:
OBJECTIVE

Primary:

To determine the effect of 5HT7 antagonism on cognition related brain activations and cognitive performance in people with bipolar disorder.

Secondary:

To examine the effect of 5HT7 antagonism on emotional processing related brain activations in people with bipolar disorder.

To examine the effect of 5HT7 antagonism on behavioral measures of mood.

Exploratory:

To determine whether early behavioural 5HT7 antagonist drug effects can be detected which may be linked to altered brain activations.

To explore whether factors, such as baseline measures of cognitive impairment and polygenic risk score, predict the extent of JNJ-18038683 related treatment effects on brain activity.

STUDY DESIGN The study will use a randomized, double-blind, placebo controlled, cross-over, pharmacological functional MRI (fMRI) design to examine the neural and behavioural effects of one week's treatment with the 5HT7 antagonist, JNJ-18038683, and placebo. Participants will attend four study visits: a screening visit, a baseline visit and two neuroimaging visits. Each neuroimaging visit will be identical and comprise structural imaging, perfusion imaging with arterial spin labelling, resting state and task-based functional MRI. FMRI tasks will be working memory (N-back), emotional processing (faces), and paired associate visuospatial learning (PAL). On the neuroimaging visits, a neuropsychological battery will also be performed, subjective and behavioural effects will be assessed with standard questionnaires and adverse events will be recorded.

NUMBER OF SUBJECTS 34 cognitively impaired participants with bipolar disorder and 34 healthy participants will complete the study. Replacements are allowed in case of drop-out.

TARGET POPULATION Male and female patients with a current diagnosis of Bipolar Disorder and healthy volunteers. All participants will be right-handed. Patients will be primarily recruited through South London and Maudsley NHS Foundation Trust clinical services, with other trusts potentially contributing to recruitment. Participants will also be recruited by public advertising, online and social media and through NIHR Mental Health CRN. Healthy volunteers will be recruited through advertisement within King's College London, in the local press, online and through contacting participants from previous studies who have expressed an interest in further research participation.

STUDY DRUG (DOSE/ROUTE/REGIMEN) Name of product: JNJ-18038683, an investigational drug, a 5HT7 antagonist Dose: 20mg once daily Administration: Oral Duration of dosing: One week

JNJ-18038683 and matching placebos will be provided by Janssen Research and Development, LLC, the manufacturer of JNJ-18038683.

ASSESSMENTS:

Screening visit (Visit 1):

Participant's cognitive; mood and physical health suitability will be assessed during this visit. Participants will complete the RAVLT to screen for cognitive impairment. Bipolar disorder DSM-5 diagnosis will be confirmed using the M.I.N.I. 6.0. Mood and anxiety symptoms will be assessed using the HAM-D, YMRS, QIDS-CR, C-SSRS, Altman Self-Rating Mania scale and HAM-A mood rating scales. Substance use will be assessed using the cannabis experiences, Fagerstrom smoking and AUDIT alcohol questionnaires. All participants will undergo a physical examination, ECG, urine drug screen, breath alcohol test, pregnancy test for females, urinalysis and blood will be taken to assess hepatic, renal and haematological function and to determine bipolar disorder polygenic risk scores.

Baseline visit (Visit 2) If the screening assessments indicate suitability, participants will then attend a baseline visit. They will complete a brief physical health examination including recording vital signs, ECG, urine drug screen, breath alcohol test and a pregnancy test for females. Mood and anxiety symptoms will be assessed using the HAM-D, YMRS, QIDS-CR, C-SSRS, Altman Self-Rating Mania scale and HAM-A mood rating scales. Sleep will be assessed using the PSQI. Cognition will be assessed using the ISBD-BANC cognitive battery and subjective cognitive impairment will be assessed using the PDQ and FAST questionnaires. Participants will be provided with the week 1 study medication pack, determined by randomization code, and a study diary to record taking each day's medication and any adverse events experienced.

Imaging visits (Visit's 3 and 4):

Participants will undergo a brief medical examination, ECG and urine drug screen. Cognition, mood, psychosocial functioning and sleep will be assessed at each neuroimaging visit using the ISBD-BANC, PDQ, QIDS-CR, C-SSRS, YMRS, FAST and PSQI. A blood sample will be taken at each visit to monitor hepatic, renal and haematological functions and so that plasma can be stored to potentially measure JNJ-18038683 levels. During each imaging session, participants will complete the n-back working memory, paired associate visuospatial learning (PAL), and emotional faces recognition fMRI tasks, an arterial spin labelling (ASL) scan to assess cerebral blood flow, a resting state scan, and a T1 and T2 structural scan.

PROCEDURES

Randomisation:

Participants will be randomized into the study provided they have satisfied all selection criteria. Each participant will be assigned to a sequence of treatment administrations by means of a computer-generated, pseudo random code based on stacks of William's Squares, to ensure each treatment is equally distributed across each study period. A blinded randomization list will be provided by the pharmacist or delegate to the investigator and, in accordance with the randomization list, if a participant is withdrawn from the study, the replacement participant will be allocated to the same treatment sequence as the subject they are replacing. Replacement numbers will be discussed and agreed between the investigator and the pharmacist.

Analytical Plan:

A brief plan for data analysis is provided in the main body of the protocol. A detailed Statistical Analytical Plan will be produced before the end of the data collection phase of the study. A brief description of the main endpoints is provided here:

Primary endpoints:

1. Change in cognitive task related right superior frontal gyrus and dorsolateral prefrontal cortex brain activations associated with JNJ-18038683 treatment.
2. Change in cognitive performance, as measured by change in International Society for Bipolar Disorders Battery for the Assessment of Cognition (ISBD-BANC) test battery composite score, associated with JNJ-18038683 treatment (Co-primary).

Secondary endpoints:

1. Change in emotional processing related amygdala brain activations associated with JNJ-18038683 treatment.
2. Change in cognitive and emotional network connectivity associated with JNJ-18038683 treatment.
3. Change in other behavioural measures of cognition (ISBD-BANC test battery individual task scores) and mood scores (Quick Inventory of Depressive Symptomatology, Young Mania Rating Scale) associated with JNJ-18038683 treatment.

Safety:

Listings, summary tables and graphs will be produced for safety and tolerability assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handed participants between the ages of 18 and 60 years, inclusive, who are currently in a euthymic mood state defined as ≤8 on the Hamilton Rating Scale for Depression (HAM-D) and Young Mania Rating Scale (YMRS).
2. The participant has a resting pulse ≥51 bpm and ≤100 bpm.
3. The subject has a resting systolic blood pressure ≥91 mmHg and ≤140 mmHg and a resting diastolic blood pressure ≥51 mmHg and ≤90 mmHg at the Screening Visit. An out-of-range resting systolic blood pressure may be repeated if a medically valid reason is present, for example, the subject suffers from white-coat hypertension or experienced stress (e.g. late arrival).The medically valid reason must be documented and signed by the investigator.
4. The subject has clinical laboratory test values within the reference ranges based on the blood and urine samples taken at the Screening Visit. Borderline value parameters may be accepted if they are, in the opinion of the investigator, clinically insignificant.
5. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
7. Ability to understand written and verbal instructions in English.
8. Women of child bearing potential must have a negative pregnancy test at screening and at baseline visits and must agree to use a medically accepted method of contraception throughout the study.

Exclusion Criteria:

1. Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing), and any primary psychiatric diagnosis other than bipolar disorder.
2. Participants who have used or plan to use during the conduct of the study:

   1. Fluoxetine within 5 weeks prior to the baseline visit or during the study
   2. Monoamine oxidase inhibitors within 3 weeks of the baseline visit or during the study
   3. Other prescription medication within 7 days prior to the baseline visit or within or 5 half-lives (whichever is longer) with the exception of the following which are allowed:

   i. For the bipolar disorder group, prescribed psychotropic medications as long as they are not included in the list of CYP2D6 and CYP2C19 medications listed in exclusion's 3 and 4 below.

   ii. Limited use (not more than 3 days per week) medications (non CYP2D6 or CYP2C19 substrates) such as prn treatments for asthma or acute migraine.

   iii. Women who are taking hormone replacement therapy or hormonal contraception must be on a stable regimen for 30 days prior to screening and remain on that regimen throughout the study

   iv. Paracetamol may be used at doses of 1 g/day

   Herbal supplements must be discontinued 28 days prior to the first dose of study medications. At the discretion of the investigator a shorter drug free or discontinuation period may be acceptable depending on the precise drugs/supplements taken.
3. As JNJ-18038683 is a strong inhibitor of cytochrome P450 2D6, use of the following CYP2D6 substrates will be an exclusion: carvedilol, S-metoprolol, propafenone, timolol, amitriptyline, clomipramine, desipramine, fluoxetine, imipramine, paroxetine, venlafaxine, haloperidol, perphenazine, risperidone, thioridazine, zuclopenthixol, alprenolol, amphetamine, aripiprazole, atomoxetine, bufuralol, chlorpheniramine, chlorpromazine, clonidine, codeine, debrisoquine, dexflenfluramine, dextromethorphan, donepezil, duloxetine, encainide, flecainide, fluvoxamine, lidocaine, metoclopramide, methoxyamphetamine, mexilletine, minaprine, nebivolol, nortriptyline, ondansetron, oxycodone, perhexiline, phenacetin, phenformin, promethazine, propafenone, propranolol, sparteine, tamoxifen, tramadol, venlafaxine. Participants planning to use these medications after their participation in the study must commit to a two-week washout period at the end of the study before commencing these medications.
4. As JNJ-18038683 is a moderate inhibitor of cytochrome P450 2C19, use of the following CYP2C19 substrates will be an exclusion: Proton pump inhibitors, phenytoin, phenobarbitone, diazepam, Norphenytoin, S-mephenytoin, phenobarbitone, amitriptyline, carisoprodol, citalopram, chloramphenicol, clomipramine, clopidogrel, cyclophosphamide, hexobarbital, imipramine, indomethacin, labetalol, R-mephobarbital, moclobemide, nelfinavir, nilutamide, primidone, progesterone, proguanil, propranolol, teniposide, warfarin, voriconazole. Participants planning to use these medications after their participation in the study must commit to a two-week washout period at the end of the study before commencing these medications.
5. Currently taking medications with significant 5HT7 antagonist properties (eg lurasidone, vortioxetine)
6. Treatment with another experimental medicine drug within the 3 months preceding the first dose of study medication, over the course of the study, and two weeks after discontinuing study medications
7. History of sensitivity to JNJ-18038683 or other medications with 5HT7 antagonist properties.
8. History of febrile illness within 5 days prior to the first dose.
9. Any condition possibly affecting drug absorption (eg, gastrectomy).
10. 12-lead ECG considered abnormal by a clinician
11. A positive urine drug screen on or after the screening visit during their active involvement in the study for opiates, methadone, cocaine, amphetamines (including MDMA), barbiturates, benzodiazepines and cannabinoids.
12. Unwilling or unable to comply with the Lifestyle guidelines.
13. Participants who, in the opinion of the investigator, have any medical or psychological condition or social circumstances which would impair their ability to participate reliably in the study, or who may increase the risk to themselves or others by participating.
14. Diagnosis of alcohol or drug dependence in the year prior to recruitment or diagnosis of harmful use of alcohol or drugs within the previous 6 months.
15. Female participants of child bearing potential who are not using adequate contraception as specified in above criteria for inclusion.
16. Female participants that are currently pregnant or are breast feeding.
17. A history of moderate to severe head injury or neurological conditions that may impair cognitive performance
18. Ineligibility to undergo MRI imaging, for example the presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies as assessed by a standard pre-MRI questionnaire.
19. Participant weight in excess of 126kg or physical dimensions such that the participant may not fit in the MRI scanner.
20. A history of claustrophobia or participant feels unable to lie in a MRI scanner for a period of around one hour.

Additional exclusion criteria for participants with bipolar disorder

1. Significant change in dose or type of prescribed psychotropic medications in the month prior to the Screening visit or likely change during the study.

Additional exclusion criteria for healthy participants

1. A personal history of any significant psychiatric disorder including a history of suicide attempts or significant suicidal ideation or a family history of severe mental illness (such as psychosis, bipolar disorder or schizophrenia).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
fMRI imaging | after 7 days on either placebo or JNJ-18038683
  Change in cognitive task related right superior frontal gyrus and dorsolateral prefrontal cortex brain activations associated with JNJ-18038683 treatment.
ISBD-BANC | after 7 days on either placebo or JNJ-18038683
  Change in cognitive performance, as measured by change in International Society for Bipolar Disorders Battery for the Assessment of Cognition (ISBD-BANC) test battery composite score, associated with JNJ-18038683 treatment

SECONDARY OUTCOMES:
fMRI imaging | 7 days
  Change in emotional processing related amygdala brain activations associated with JNJ-18038683 treatment.
fMRI imaging | 7 days
  Change in cognitive and emotional network connectivity associated with JNJ-18038683 treatment.
QIDS-CR - Quick Inventory of Depression Symptomology | 7 days
  Change in mood associated with JNJ-18038683 treatment.
YMRS - Young Mania Rating Scale | 7 days
  Change in mood associated with JNJ-18038683 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stokes, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom